CLINICAL TRIAL: NCT01466049
Title: Evaluation of New Biomarker Assays in Ovarian Cancer Patients Presenting to a Generalist With an Adnexal Mass
Brief Title: New Biomarkers Evaluating Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-35
Record Dates: First submitted 2011-11-03; First posted 2011-11-07 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Adnexal Mass
Keywords: Ovarian Cancer; Adnexal Mass; Pelvic Mass
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate new biomarkers for patients presenting to a physician for surgery to remove a mass in their pelvis and to continue to evaluate these types of patients using the ROMA algorithm for post-market benefits.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years or older
* Adnexal mass present documented by imaging
* Scheduled to undergo surgery based on a finding of adnexal mass
* Able and willing to provide Informed Consent

Exclusion Criteria:

* Previous history of ovarian cancer
* Previous history of bilateral oophorectomy
* Currently known to be pregnant
* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with an adnexal mass, presenting to a general surgeon or obstetrician/ gynecologist at a general or specialty center within the United States, for whom a decision to proceed with surgery to remove the mass has been made.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluate novel biomarkers for patients with an adnexal mass | observational studies

CONTACTS AND LOCATIONS:
Overall Officials: Diana Dickson, Study Director — Fujirebio Diagnostics, Inc.
Locations (2):
- United States (2):
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma